CLINICAL TRIAL: NCT06900283
Title: Quality of Life as a Predictor of Mortality and Progression-free Survival in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Quality of Life as a Predictor of OS and PFS in Patients With Lung Cancer
Acronym: FACT-L_Pred
Status: Active, not recruiting | Type: Observational
Sponsor: Instituto Nacional de Cancerologia, Columbia (Other Government)
Collaborators: Hospital Universitario San Ignacio (Other); Hospital Pablo Tobón Uribe (Other); Hospital Alma Mater de Antioquia (Unknown)
Responsible Party: Sponsor
Other Study IDs: C19010300492 - FACT-L; C19010300492 (Other: Instituto Nacional de Cancerología)
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancers; Lung Cancer, Non-Small Cell
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
By 2020, lung cancer continues leading the first cause of cancer mortality and the second most common type of cancer in the world. There are limitations to early detection and then more than 60% of patients are diagnosed in advanced stages where there are no longer curative options; that situation is associated with high mortality and poor survival. It is known that some clinical and biochemical parameters of the disease have been recognized as prognostic factors; however, it has been described that a reduction in the overall global quality of life score, mainly by physical function, increased pain, and dysphagia, are associated with mortality, and having high social well-being and global quality of life scores are associated with a lower risk of death.

Objective: This study will measure association between Health-Related Quality of Life levels and mortality and progression free survival in advanced non-small cell lung cancer patients

Patients and methods:

This study will include patients with lung cancer histopathological confirmed including bronchus or trachea.

Methodologically, the study has two components: One related to the exposure variable (HRQL), which involves a scale validation study, and other related to the measurement of the association between HRQoL and survival outcomes, which involves a prospective cohort analytical observational study. This last component will be carried out specifically with a sample of patients with non-small cell lung cancer (NSCLC).

Results and impact: The project contribute to the implementation of tools adapted and validated in the Colombian context to assess the quality of life in patients with lung cancer. Additionally, knowing the relationship between quality of life and traditional oncological outcomes will provide tools to give patients with comprehensive treatment, and to have a prognosis of the disease that incorporates psychosocial aspects

DETAILED DESCRIPTION:
The validation process of the scale includes the evaluation of internal consistency, content validity, sensitivity to change, test-retest reliability and the data will be analyzed according to the item response theory. In the cohort study, the association between HRQoL levels, mortality and progression-free survival will be measured in 250 patients with non-small cell lung cancer.

Analysis plan: Conventional methods of descriptive statistics will be applied in accordance with the characteristics of the variables. For validation procedures, exploratory and confirmatory factorial analysis techniques, estimation of correlation and internal consistency coefficients, and methods to compare means in repeated measures (ANOVA of repeated measures) will be used. In the cohort study, time-to-event models will be used (Cox proportional hazards models or parametric models, depending on the fulfillment of assumptions). Since the independent variable will have different times of measurement, time-to-event models will include methods that handle covariates that change over time.

ELIGIBILITY:
Inclusion Criteria:

1. Have a confirmed histologic diagnosis of non-small cell lung cancer
2. Advanced stage (III to IV)
3. 8 years older
4. Voluntary acceptance of participation

Exclusion Criteria:

1. Present cognitive or sensory deficits that make it difficult to process the instruments used in the research
2. Metachronous tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced lung cancer
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 36 months
  Overall survival (OS) is the average amount of time a patient survives after being diagnosed with or starting treatment for a disease

SECONDARY OUTCOMES:
Disease-Free Survival (DFS) | 36 months
  Disease-free survival (DFS) is the time after treatment when a patient is free of cancer signs and symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Carreno, Md, Principal Investigator — Instituto Nacional de Cancerologia, Columbia
Locations (1):
- Instituto Nacional de Cancerologia, Bogota, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No